CLINICAL TRIAL: NCT03212755
Title: Serum Immunoglobulin (G ) as a Predictive Marker of Early Renal Affection in Type 2 Diabetic Patients
Brief Title: Serum Immunoglobulin (G) as a Marker of Diabetic Nephropathy
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Seham Mohammed Ali, principal investigator, Assiut University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Screening
Other Study IDs: PRUD
Record Dates: First submitted 2017-07-07; First posted 2017-07-11 (Actual); Last update posted 2017-07-11 (Actual); Status verified 2017-07

CONDITIONS: Diabetic Nephropathies
MeSH Terms: conditions — Diabetic Nephropathies

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- group 1 (Experimental): 25 diabetic patients without diabetic nephropathy
  Interventions: Diagnostic Test: serum immunoglobulin G level
- group 2 (Experimental): 25 type 2 diabetic patients with diabetic nephropathy
  Interventions: Diagnostic Test: serum immunoglobulin G level
- group 3 (Sham Comparator): 25 healthy subjects
  Interventions: Diagnostic Test: serum immunoglobulin G level

INTERVENTIONS:
Diagnostic Test: serum immunoglobulin G level — measurement of the serum level as a marker of diabetic complications

SUMMARY:
Diabetes mellitus is a chronic disease that affects 366 million people worldwide ( 6.4 % of the adult population ) and is expected to rise to 522 million by 2030 . Diabetic nephropathy occurs in approximately one - third of all people with diabetes and is the leading cause of renal failure in developed and developing countries Diabetic nephropathy is a severe complication occurring in diabetic patients and it is associated with an increased risk of all- cause mortality , cardiovascular disease and progression to end stage renal disease , requiring costly renal replacement therapy in the form of dialysis or transplantation

ELIGIBILITY:
Inclusion Criteria:

* type 2 diabetic patients

Exclusion Criteria:

* patients with diabetes type 1 ,
* pregnant and lactating females ,
* patients with any congenital disease , Infection , Smokers , alcoholics , and drug abusers .

Ages: 30 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 75 (Estimated)
Dates: Start 2017-08 (Estimated); Primary Completion 2019-06 (Estimated); Study Completion 2019-12 (Estimated)

PRIMARY OUTCOMES:
The number of patients with high level of immunoglobulin in serum | 24 hours

IPD SHARING:
Plan to Share IPD: No